CLINICAL TRIAL: NCT06685588
Title: Efficacy of Topical 5-FUvs Calcipotriol As PDT Pre-treatment for Field Actinic Keratoses
Brief Title: Efficacy of Topical 5-Fluorouracil Vs Calcipotriol As Photodynamic Therapy Pre-treatment for Field Actinic Keratoses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Maeve Herlihy, Dr Maeve Herlihy, St Vincent's University Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RS24-046
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Actinic Keratosis of Face and Scalp; Actinic Keratoses
Keywords: efudix; dovonex; 5-fluorouracil; calcipotriol; actinic keratosis; actinic keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil; calcipotriene

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Calcipotriol / Dovonex (Active Comparator): Randomised to PDT pre-treatment with calcipotriol
  Interventions: Drug: 5-FU (fluorouracil); Drug: Calcipotriol
- Calcipotriol /Dovonex (Active Comparator): Calcipotriol pre-treatment prior to PDT
  Interventions: Drug: 5-FU (fluorouracil); Drug: Calcipotriol

INTERVENTIONS:
Drug: 5-FU (fluorouracil) — Topical 5-FU (fluorouracil) pretreatment prior to dovonex
  Other Names: Efudix
Drug: Calcipotriol — Calcipotriol pre-treatment prior to PDT

SUMMARY:
The purpose of this study is to compare two different creams (5-fluorouracil, known as Efudix, and calcipotriol, known as Dovonex) to see which one works better when used before Photodynamic Therapy (PDT) to treat sun-damaged skin on the scalp (called actinic keratoses).

PDT is often used on its own to treat these spots, but it doesn't always remove them completely. Using Efudix or Dovonex before PDT might improve the results, but we don't yet know which is better.

The main questions are -

1. Is efudix or dovonex better at treating actinic keratoses when used prior to PDT
2. Is efudix or dovonex more tolerable for patients?

Participants will be randomised to treat their scalp with efudix or dovonex for seven days prior to their first PDT treatment. They will be reviewed on day 7, prior to starting PDT, and again a week later when they present for their second PDT treatment.

During follow up, patients will be reviewed at 28 days, 3, 6, 9, and 12 months after treatment.

At each of these visits, the number of actinic keratoses will be counted, graded, mapped and photographed to allow assessment of improvement before and after treatment.

DETAILED DESCRIPTION:
1. Recruitment We will enrol 50 number of patients in our department who have been referred for daylight PDT treatment of actinic keratoses on the scalp and forehead. The patients will be given a study specific number based on the order of their enrolment. 25 patients will be randomised to be pre-treated with calcipotriol and 25 with 5-FU.
2. Demographic data recorded Relevant baseline characteristics will be registered at baseline visit (prior history of skin cancer, smoking yes/no, history of sun exposure, use of immunosuppressant medication in history, prior treatments for AK.
3. Initial visit - counting AKs / mapping / photos The boundaries of the area to be treated will be defined and marked using a skin marker. Photographs will be taken of right and left scalp, and the scalp straight on - with the study number and markings visible.

   We will count the AKs in each treatment area, then grade, mark and map them. AKs will be graded using the Olsen classification system. Grade 1 means they are hardly visible but palpable. Grade 2 means they are visible and palpable. Grade 3 means they are hyperkeratotic. We will photograph the treatment areas again as outlined above, with the AKs marked.

   In all patients hyperkeratotic lesions will be pre-treated with paraffin gel to remove keratotic debris. Photographs will be taken as above with the AKs marked using a skin marker.

   A polythene map will be made by marking over each previously marked AK and the outline of template, marked with surface landmarks for purpose of locating treatment site at follow-up. This will be photographed as above.
4. Randomisation & Blinding Randomisation will be achieved by block randomisation (1:1) with the patient choosing an envelope with a card marked 5-FU or calcipotriol, which will determine which pre-treatment is used.

   The phototherapy nurses will be unblinded and will apply the pre-treatments. Investigators MH, BM and AL will all be blinded to which treatment the patient is for patient reviews.
5. Pre-treatment Initially, patients will present to the department for pre-treatment. Prior to pre-treatment, the treatment will be marked out using the patients previous photos and polythene maps as a reference.

   A thin layer of the assigned pre-treatment will be applied to the patients scalp.

   On the first day of pre-treatment, it will be applied by the dermatology nurses who will educate the patient (+/- a family member) on how to apply. A new tube of the assigned pre-treatment will be opened for each patient, and they will be given this to take home. The patient (or a family member) can apply the next six days of pre-treatment themselves at home - in the same way, applying a thin layer to cover the whole treatment area once a day, at the same time each day.

   Patients will be instructed to attend for PDT treatment the day after finishing pre-treatment and for a second PDT treatment a week later.
6. PDT treatment One week after starting pre-treatment, patients will be brought in for treatment with daylight PDT. Approximately 1 gram of MAL cream will be applied on the treatment area and the area will be occluded. After a half hour the occlusive dressing will be removed and the area will be treated with a VTAC LED Floodlight SMD SAMSUNG Chip Slim Black Body 4000K (white light). The flood lamp will be orientated to provide uniform power distribution across the treatment area. White light irradiance will be measured at treatment site prior to commencement of treatment to ensure optimised setup. Patients and staff will be provided with a visor and googles for eye protection and monitored with a camera in case they become unwell while receiving treatment. It is anticipated they will receive a dose equivalent to spending two hours outside on an overcast day.

   The White light source will be commissioned and tested by Medical Physicists (JMcC / EL) in advance of the therapy. The spectral light output, light distribution, stability and uniformity will be assessed.

   The patient will rate their pain using visual analogue score (VAS) (1-100) at 1, 30, 60, 90 and 120 minutes for both treatments. To use this the patient will move a counter along 100mm scale from "no pain" to "worst pain ever". The flip side of the scale indicates the score numerically. Our nurses will record the numerical pain score and patients will not be aware of this value. If treatment has to be discontinued because of pain the timing of this will be recorded.

   Any adverse events will be recorded including erythema (mild/moderate/severe), erosions (mild/moderate/severe), pain rated out of 100 with a visual analogue score, duration of any pain and any unexpected adverse events that occur. Patients will be reviewed at 1 and 7 days following treatment for adverse events. Patients will be assessed by one investigator (MH) for local reactions such as erythema and erosions and asked to indicate how long pain persisted.

   The treatment will be repeated a week later. Again patients will rate their pain using VAS and any adverse events recorded as outlined above.
7. Study Assessments To assess clinical response, patients will be assessed 28 days after their last PDT treatment by a second investigator (AL / BM). This investigator will be blinded as to which pre-treatment modality was used for which treatment field. She will record if the patient had a preference for one treatment modality. She will count, grade and map the AKs and will calculate the percentage reduction in AK count from baseline. The primary efficacy endpoint is complete clearance of AKs.

Patients will similarly be assessed at 3, 6, 9 and 12 months for clinical response.

Photographs will be taken both with and without the polythene map visible at each follow-up visit.

In case of <75% clearance of AKs at 3 months post-treatment, the same treatment will be repeated. This will be recorded. Lesions that need additional treatment (e.g. cryosurgery, biopsy) are evaluated as non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years old)
* Field actinic keratoses on scalp
* Generally good health

Exclusion Criteria:

* Immunosuppression
* Unable to provide consent
* Abnormal photosensitivity
* Contact allergy to metvix / 5-FU / calcipotriol / topical corticosteroids
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment as assessed by proportion of participants with complete clearance of AKs from baseline (100% reduction) | 6 months post treatment
  Assessed by number of participants with complete clearance of AKs at 6 months post treatment. Complete clearance is is defined as 100% reduction in the number of AKs from baseline. AKs will be counted, marked, mapped and photographed at each visit.
Tolerability of treatment | Day of treatment, day 7 and day 28
  assessed by pain scores (visual analogue scale, 0-10), documentation of local effects such as erythema and erosions and recording of any adverse events

SECONDARY OUTCOMES:
Near-complete response | 3, 6, 9 and 12 months post treatment
  number of participants with ≥ 75% reduction in number of AK lesions
Partial response rate | 3, 6, 9 and 12 months post treatment
  number of participants with 50-75% reduction in number of AK lesions
Treatment failure rate | 3, 6, 9 and 12 months post treatment
  number of participants treatment with <50% reduction in number of AK lesions
Decrease in number AK from baseline per patient | 1, 3, 6, 9 and 12 months post final treatment.
Proportion of patients who develop a SCC in the treatment area during study follow-up period | 12 months
Complete response at 3,9 & 12 months | 3, 9 and 12 months post treatment
  number of participants with 100% clearance as measured at 3,9 & 12 months. Primary outcome measure is complete clearance at 6 months.

IPD SHARING:
Plan to Share IPD: No